CLINICAL TRIAL: NCT01874912
Title: Human Irisin Concentration in Sarcopenia
Status: Completed | Type: Observational
Sponsor: Korea University (Other)
Responsible Party: Principal Investigator, K. M. Choi, Professor, Korea University
Other Study IDs: SO(IRISIN)
Record Dates: First submitted 2013-06-03; First posted 2013-06-11 (Estimated); Last update posted 2013-06-11 (Estimated); Status verified 2013-06

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Irisin has been identified as a novel myokine that drives brown-fat-like conversion of white adipose tissue. In this cross-sectional study, the researches investigated whether serum irisin levels are decreased in patients with sarcopenia compared with control subjects with normal muscle mass, and assessed the association between serum irisin levels and various metabolic parameters.

ELIGIBILITY:
Inclusion Criteria:

* 20<age<80
* apparently healthy subjects

Exclusion Criteria:

* a history of cardiovascular disease
* diabetes
* stage 2 hypertension
* malignancy
* severe renal or hepatic disease

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients in Korean Sarcopenic Obesity Study (KSOS), an prospective observational cohort study designed to examine the prevalence of sarcopenia and sarcopenic obesity in Korean adults and to evaluate their effects on metabolic disorders and health outcomes.
Sampling Method: Probability Sample
Enrollment: 406 (Actual)
Dates: Start 2009-11; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Serum concentration of irisin in the subjects with sarcopenia | 12 week

SECONDARY OUTCOMES:
The relationship of serum irisin levels with lipid profiles | 12 week
The relationship of serum irisin levels with skeletal muscle mass index | 12 wks

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Guro Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Choi HY, Kim S, Park JW, Lee NS, Hwang SY, Huh JY, Hong HC, Yoo HJ, Baik SH, Youn BS, Mantzoros CS, Choi KM. Implication of circulating irisin levels with brown adipose tissue and sarcopenia in humans. J Clin Endocrinol Metab. 2014 Aug;99(8):2778-85. doi: 10.1210/jc.2014-1195. Epub 2014 Apr 29. PMID 24780049